CLINICAL TRIAL: NCT03236701
Title: The Impact of a Nutritional Intervention Based on Egg White for Phosphorus Control in Haemodialysis Patients
Brief Title: Egg White for Phosphorus Control in Haemodialysis Patients
Acronym: UAUDIPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruna Guida, Associate Professor in Physiology, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76/17
Record Dates: First submitted 2017-07-24; First posted 2017-08-02 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Renal Insufficiency, Chronic; Dialysis; Hyperphosphatemia
Keywords: hyperphosphatemia; hemodialysis; dietary treatment; egg white; protein energy wasting
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): usual diet
- Intervention (Experimental): egg white instead of meat or fish in two meals twice a week for three months
  Interventions: Other: Egg White replacement

INTERVENTIONS:
Other: Egg White replacement — Nutritional intervention: the meat or fish of two meals will be replaced twice a week with an equivalent amount (in protein content) of egg white.
  Arms: Intervention

SUMMARY:
To evaluate the effect on phosphatemia in hemodialysis patients of replacing the meat or fish included in two meals a week with an amount of egg white containing the same quantity of proteins.

DETAILED DESCRIPTION:
Hyperphosphatemia develops in the majority of patients with end-stage renal disease (ESRD). It is responsible for severe complications such as mineral bone disease, and has a role in worsening the cardiovascular mortality of dialyzed patients. Therefore, a close control of serum phosphorus remains a cornerstone in the clinical management of dialyzed patients to improve their long term prognosis. There are multiple sources of phosphorus in the diet that could be the target of such a dietary intervention but, because of important differences in bioavailability, they are not all equally relevant in influencing phosphatemia. Among them animal proteins that have a bioavailability of about 60% represent an important target for phosphate-lowering nutritional interventions. However, lowering the protein content of the diet in hemodialysis (HD) patients may be dangerous because it may increase the the risk of malnutrition hence worsening their prognosis. In the present study we intend to explore an alternative strategy to lower the intake of phosphate with animal proteins by replacing the meat or fish included in two meals a week with egg white that is reach of proteins but has virtually no phosphate.

ELIGIBILITY:
Inclusion Criteria:

* thrice weekly 4 h standard bicarbonate HD treatment with an at least 6-month vintage
* stable dialysis dose and modality at least by 3 months
* hyperphosphataemia (serum phosphate ≥5.0 mg/dl) at least by 3 months
* stable dietary intake at least by 3 months
* stable body weight at least by 3 months
* stable biochemical markers at least by 3 months

Exclusion Criteria:

* diabetes
* liver disease
* malignancy
* previous parathyroidectomy
* psychiatric diseases
* non-collaborative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
Decrease in serum phosphate levels | Phosphate level will be measured monthly for three months from the beginning of the study
  This is the primary outcome because of the link between cardiovascular mortality and hyperphosphatemia

SECONDARY OUTCOMES:
Changes in body composition assessed by bioelectrical impedance analysis | BIA will be performed monthly for three months from the beginning of the study
  Protein malnutrition causes a decrease in body cell mass. By bioelectrical impedance analysis (BIA) the changes in this parameter in the two experimental groups will be evaluated at one, two and three months from the beginning of the study.
Changes in serum albumin concentration | Serum albumin will be measured monthly for three months from the beginning of the study
  Protein malnutrition causes a decrease in serum albumin concentration that will be, therefore, monitored, at one, two and three months from the beginning of the study.
Changes in hemoglobin levels | hemoglobin level will be measured monthly for three months from the beginning of the study
  Protein malnutrition causes a decrease in hemoglobin levels that will be, therefore, monitored, at one, two and three months from the beginning of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University Hospital, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guida B, Parolisi S, Coco M, Ruoppo T, Veccia R, di Maro M, Trio R, Memoli A, Cataldi M. The impact of a nutritional intervention based on egg white for phosphorus control in hemodialyis patients. Nutr Metab Cardiovasc Dis. 2019 Jan;29(1):45-50. doi: 10.1016/j.numecd.2018.09.010. Epub 2018 Sep 28. PMID 30459073